CLINICAL TRIAL: NCT05160116
Title: Influence of Timing of Switch Operation in Transposition of Great Arteries
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, Department of Anesthesiology, Brugmann University Hospital
Other Study IDs: CHUB-PED-Timing_Switch
Record Dates: First submitted 2021-11-09; First posted 2021-12-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Transposition of Great Vessels
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transposition of great vessels are usually corrected by an arterial switch operation. This operation is often done during the first week of life as surgical delays lead to deconditioned left ventricle. On the other hand early surgery carries also risks as neonatal physiology may have problems adapting to an intervention under cardiopulmonary bypass, possible pulmonary hypertension. Arterial switch operation between 2008 and 2020 done at our center will be reviewed. Primary outcome will be mortality or severe postoperative morbidity. Patients will be divided in 2 groups according to the presence or absence of the primary outcome. After propensity score matching, they will be analysed according to the timing of operation.

DETAILED DESCRIPTION:
Scientific background and motivation

The transposition of great vessels (TGV) is a congenital heart defect in which the aorta follows the right ventricle and the pulmonary artery follows the left ventricle. At birth, the pulmonary and systemic circulations work in parallel and the communication between them depends on shunts in the cardiac stage (permeability of the Botal hole) or in the supra-cardiac (ducis arteriosus).

It's the most common congenital heart disease and his incidence is estimated between 0.7 and 0.8 per 1000 births. It's a pathology that may be associated with other heart defects, such as interventricular communication (IVC) or pulmonary stenosis, but rarely with a chromosomal abnormality or malformative syndrome.

TGV's manifestation is an isolated cyanosis, refractory to oxygen. And mortality reaches 90% in the first year of life in absence of treatment.

TGV's management has evolved over the last 50 years. First, thanks to the antenatal ultrasound diagnosis, allowing early strategies in postnatal to maintain a shunt between the two circulations (Prostaglandin and Balloon atrial septostomy). Then, by the evolution of corrective surgeries; indeed atrial repair techniques (Senning and Mustard) have given way to the arterial Switch with coronary reimplantation by microsurgery.

When it's possible, the operation takes place during the first week of life. Indeed, it's well established that surgical delay leads to a risk of left ventricle's deconditioned4 and sometimes impaired brain growth. But the risks of a premature surgery are less clear: Operability of the newborn, ability to tolerate an intervention under extracorporeal circulation (ECC), difficulties related to physiological pulmonary arterial hypertension at birth must be considered in the operative indication.

The ideal timing for surgery is still poorly defined. In 2014, Anderson et al showed better results for arterial Switches performed on the third day of life6. On the other hand, Kumar et al, also studied the relationship between operative timing and morbi/mortality of several congenital heart surgeries including the arterial Switch but they found no relationship between them.

Study design

The investigators would like to establish if there is a relationship between the age of the newborn at the time of surgery and postoperative morbi/mortality. Therefore, the investigators want to review all the medical records of children operated on a TGV by the arterial Switch technique at HUDERF between 2008 and 2020. The morbidity/mortality criteria observed will be the same as those usually used in studies conducted on paediatric cardiac surgery at HUDERF:

1. The data of interest will be extracted from a database built up over years summing up the medical records of cardiac operated patients since 2002.
2. Statistics:

2.1. Children will be divided into two groups according to the primary outcome (present or absent). They will be matched using a propensity analysis and then compared in terms of operating time.

2.2. The influence of operative time on the occurrence of the primary outcome will also be analysed by a linear regression technique in which the parameter "operating time" will be considered as a continuous variable.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with TGV and
* operated at HUDERF between 2008 and 2020 and
* arterial switch operation

Exclusion Criteria:

* Any surgical technique other than the switch operation for TGV
* patients operated before 2008

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children with TGV operated by an arterial switch operation between 2008 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Mortality | From operation until 28 days postoperatively
  death (percent) during hospitalization
Incidence (percent) of severe postoperative morbidity | From operation until 28 days postoperatively
  Severe postoperatively morbidity is defined as patients meeting at least 2 of the following events:
  * respiratory failure defined as duration of mechanical ventilation > 75th percentile of our cohort
  * prolonged inotropic support defined as duration of inotropic support > 48 hours
  * renal failure defined as glomerular filtration rate (GFR) decreased more than 75% compared to preoperative GFR
  Every patient meeting at least 2 of these 3 events will be counted as having severe postoperative morbidity.
  Total incidence (expressed as percent of total population) of severe postoperative morbidity will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — Brugmann University Hospital & HUDERF
Locations (1):
- Hôpital Universitaire des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagata H, Glick L, Lougheed J, Grattan M, Mondal T, Thakur V, Schwartz SM, Jaeggi E. Prenatal Diagnosis of Transposition of the Great Arteries Reduces Postnatal Mortality: A Population-Based Study. Can J Cardiol. 2020 Oct;36(10):1592-1597. doi: 10.1016/j.cjca.2020.01.010. Epub 2020 Jan 20. PMID 32622839
- [Background] Sidi D, Planche C, Kachaner J, Bruniaux J, Villain E, le Bidois J, Piechaud JF, Lacour-Gayet F. Anatomic correction of simple transposition of the great arteries in 50 neonates. Circulation. 1987 Feb;75(2):429-35. doi: 10.1161/01.cir.75.2.429. PMID 3802447
- [Background] Lim JM, Porayette P, Marini D, Chau V, Au-Young SH, Saini A, Ly LG, Blaser S, Shroff M, Branson HM, Sananes R, Hickey EJ, Gaynor JW, Van Arsdell G, Miller SP, Seed M. Associations Between Age at Arterial Switch Operation, Brain Growth, and Development in Infants With Transposition of the Great Arteries. Circulation. 2019 Jun 11;139(24):2728-2738. doi: 10.1161/CIRCULATIONAHA.118.037495. Epub 2019 May 28. PMID 31132861
- [Background] Anderson BR, Ciarleglio AJ, Hayes DA, Quaegebeur JM, Vincent JA, Bacha EA. Earlier arterial switch operation improves outcomes and reduces costs for neonates with transposition of the great arteries. J Am Coll Cardiol. 2014 Feb 11;63(5):481-7. doi: 10.1016/j.jacc.2013.08.1645. Epub 2013 Oct 30. PMID 24184243
- [Background] Kumar TK, Charpie JR, Ohye RG, Hirsch-Romano JC, Donohue JE, Yu S, Sood V, Wilkinson DA, Nelson K, Mitchell E, Goldberg CS, Gaies MG. Timing of neonatal cardiac surgery is not associated with perioperative outcomes. J Thorac Cardiovasc Surg. 2014 May;147(5):1573-9. doi: 10.1016/j.jtcvs.2013.07.020. Epub 2013 Aug 26. PMID 23988282
- [Background] Willems A, Datoussaid D, Tucci M, Sanchez Torres C, De Ville A, Fils JF, Van der Linden P. Impact of On-Bypass Red Blood Cell Transfusion on Severe Postoperative Morbidity or Mortality in Children. Anesth Analg. 2016 Aug;123(2):420-9. doi: 10.1213/ANE.0000000000001425. PMID 27331784